CLINICAL TRIAL: NCT02178293
Title: MISTRAL (Mouthwash In Sore Throat Relief: Antiinflammatory vs. Local Anesthetic Therapy) "Efficacy and Tolerability of Ketoprofen Lysine Salt as a Mouthwash in Acute Phlogosis of the Pharyngeal Cavity; Multicentre, Randomized, Single-blind, Parallel-group Comparison Versus Benzidamine Hydrochloride"
Brief Title: Ketoprofen Lysine Salt as Mouthwash in Acute Phlogosis of the Pharyngeal Cavity Versus Benzidamine Hydrochloride
Acronym: MISTRAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1087.7
Record Dates: First submitted 2014-06-27; First posted 2014-06-30 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis

ARMS (2):
- Benzidamine hydrochloride (Active Comparator)
  Interventions: Drug: Benzidamine hydrochloride
- Ketoprofen lysine salt (Experimental)
  Interventions: Drug: Ketoprofen lysine salt

INTERVENTIONS:
Drug: Benzidamine hydrochloride
  Arms: Benzidamine hydrochloride
Drug: Ketoprofen lysine salt
  Arms: Ketoprofen lysine salt

SUMMARY:
A study to in order to verify any differences between the 2 treatment groups in terms of duration of analgesic effects after the first drug intake and time to remission of symptoms and signs of pharyngitis

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, aged 18 to 70 years, suffering from acute pharyngitis, pharyngolaryngitis
* Moderately or severely intense pain in the pharyngeal region (score ≥ 70 mm) from the "visual analogue scale" (VAS)
* At least 1 of the 2 inflammation signs (edema and hyperemia) to be moderately or severely intense (score ≥ 2) from the scoring scale from 0 to 3
* Release of written informed consent by the patient

Exclusion Criteria:

* Patients suffering from a microbial infection requiring specific antimicrobial treatment
* Patients who have taken the trial drugs during the week before enrolment
* Patients who have taken corticosteroids or antibiotics during the week before enrolment
* Ascertained or suspected hypersensitivity to trial drugs or to chemically correlated drugs or to other non-steroidal anti-inflammatory drugs or to mouthwashes in general
* Patients who are unable to properly fill in the diary every day as provided for by the protocol
* Ascertained or presumed pregnant or lactating women
* Inclusion in any other clinical trial during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 1998-09; Primary Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
Duration of analgesic effects in hours | Up to 6 hours

SECONDARY OUTCOMES:
Average number of days required to obtain remission of pain | Up to day 8
  day on which 2 consecutive pain measurements are both below 10 mm of the visual analog scale (VAS)
Average severity of edema and hyperemia, assessed by investigator on a 4-point-scale | Up to day 8